CLINICAL TRIAL: NCT04159818
Title: Immune Induction Strategies to Improve Response to Immune Checkpoint Blockade in Triple Negative Breast Cancer (TNBC) Patients: the TONIC-2 Trial
Brief Title: Immune Induction Strategies to Improve Response to Immune Checkpoint Blockade in Triple Negative Breast Cancer (TNBC) Patients
Acronym: TONIC-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N19TON
Record Dates: First submitted 2019-10-23; First posted 2019-11-12 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Triple negative; Metastatic disease
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Nivolumab; Cisplatin; Doxorubicin

STUDY DESIGN:
Intervention Model Description: Patients are randomized between experimental cohorts and a control cohort.
Masking Description: Patients are randomized between experimental cohorts and a control cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): no induction treatment, nivolumab 240 mg flat-dose, every 2 weeks
  Interventions: Drug: Nivolumab
- Cisplatin induction (Experimental): Cisplatin 40mg/m2, weekly for two weeks, after 2 weeks followed by nivolumab 240 mg flat-dose, every 2 weeks
  Interventions: Drug: Nivolumab; Drug: Cisplatin
- Low dose doxorubicin induction (Experimental): Low dose doxorubicin 15mg flat dose, weekly for 8 weeks, after 2 weeks followed by nivolumab 240 mg flat-dose, every 2 weeks
  Interventions: Drug: Nivolumab; Drug: Low dose doxorubicin

INTERVENTIONS:
Drug: Nivolumab — 240 mg flat-dose, every 2 weeks. From 20 weeks onwards, nivolumab will be administered every 4 weeks with a flat-dose of 480 mg starting from week 20 onwards
Drug: Cisplatin — 40mg/m2, weekly for two weeks
  Arms: Cisplatin induction
Drug: Low dose doxorubicin — 15mg flat dose, weekly for 8 weeks
  Arms: Low dose doxorubicin induction

SUMMARY:
This is a single center non-blinded randomized multi-cohort non-comparative phase II trial with a Simon's two-stage design.

DETAILED DESCRIPTION:
In the first stage, 13 evaluable patients will be accrued per cohort. Evaluable is defined as: at least one administration of nivolumab and availability of paired biopsies for immunohistochemistry (for induction treatment cohorts pre-induction and pre-nivolumab biopsies).

If there are 1 or no responses observed in these 13 patients, the cohort will be stopped. Otherwise, 21 additional patients will be accrued for a total of 34.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or incurable locally advanced triple negative breast cancer (ER < 10%, HER2 IHC 0,1+ or 2+ with no amplification)
* Metastatic lesion accessible for histological biopsy
* 18 years or older
* Maximum of three lines of chemotherapy for metastatic disease and with evidence of progression of disease. Treatment with low-dose doxorubicin in the palliative setting is not allowed.
* WHO performance status of 0 or 1
* Measurable or evaluable disease according to RECIST 1.1
* Disease Free Interval (defined as time between first diagnosis or locoregional recurrence and first metastasis) longer than 1 year
* Subjects with brain metastases are eligible if these are not symptomatic and free of progression of at least 4 weeks
* A maximum dosage of 360 mg/m2 of anthracyclines and no previous anthracycline-related cardiac toxicity. In case of radiation in the cardiac area, hypertension, diabetes mellitus or hypercholesterolemia, the left ventricular ejection fraction must be 50% or higher.
* Adequate bone marrow, kidney and liver function

Exclusion Criteria:

* uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris
* known history of leptomeningeal disease localization
* history of having received other anticancer therapies within 2 weeks of start of the study drug
* history of immunodeficiency, autoimmune disease, conditions requiring immunosuppression (>10 mgl daily prednisone equivalents) or chronic infections.
* prior treatment with immune checkpoint inhibitors.
* active other cancer
* history of uncontrolled serious medical or psychiatric illness
* current pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | assessed monthly until progression or date of death; median 12 months
  Time from randomization to date of first tumor progression

SECONDARY OUTCOMES:
Overall response rate | assessed at week 6, 12 and 20 and every 8 weeks thereafter; assessed up to 120 months
  complete response or partial response according to iRECIST and RECIST1.1
Clinical benefit rate | assessed at week 6, 12 and 20 and every 8 weeks thereafter; assessed up to 120 months
  Beneficial response (complete response, partial response or stable disease) according to RECIST 1.1 and iRECIST
Overall survival | assessed monthly until date of death; median 12 months
  time from nivolumab initiation to death from any cause
Toxicity of all study regimens | assessed until 100 days after of treatment end
  adverse events will be graded according to NCI Common Toxicity Criteria v 5.0
Progression Free Survival after 6 cycles | time from nivolumab initiation to tumor progression or death from any cause; assessed up to 120 months
  the number of patients free of progression after 6 cycles of nivolumab

CONTACTS AND LOCATIONS:
Overall Officials: Marleen Kok, MD, Principal Investigator — NKI-AvL
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands